CLINICAL TRIAL: NCT00908024
Title: A Phase I/II Trial of BMS-754807 in Combination With Cetuximab (Erbitux®) in Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Combination Study of BMS-754807 and Erbitux® in Subjects With Advanced or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA191-006; EUDRACT: 2009-013766-78
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Cancer; Head and Neck Cancer; Neoplasm Metastasis
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Neoplasm Metastasis | interventions — BMS 754807; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-754807 + cetuximab (Experimental): Combination
  Interventions: Drug: BMS-754807; Drug: cetuximab (Erbitux®)

INTERVENTIONS:
Drug: BMS-754807 — Tablets, Oral, doses vary during dose escalation, once daily, varies - treatment is continued to disease progression or MD/subject/sponsor decision
Drug: cetuximab (Erbitux®) — IV infusion, IV, 400 mg/m² loading dose, then 250 mg/m², weekly, varies - treatment is continued to disease progression or MD/subject/sponsor decision
  Other Names: Eributux®

SUMMARY:
The study is expected to identify a safe dose of BMS-754807 to be given in combination with a standard dose of cetuximab and the recommended dose or dose range for Phase II studies. The study is also intended to collect first data on the effects of the combination of BMS-754807 with cetuximab on tumors of patients with colorectal cancer or squamous cell cancer of the head and neck for whom cetuximab-containing therapies have not been effective

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* ECOG status 0 - 1
* Dose escalation: Subjects with locally advanced or metastatic solid tumors who are eligible to receive cetuximab treatment and have archived tumor biopsy material available. Colorectal cancer subjects must be confirmed KRAS wild type
* Dose expansion: CRC (KRAS-WT) and head & neck cancer subjects only

  1. must be able to provide 2 fresh tumor biopsy samples
  2. must have failed one prior cetuximab-containing treatment

Exclusion Criteria:

* Symptomatic brain metastasis
* Prior treatments with anti-EGFR (except cetuximab) or anti-IGF-1R agents, experimental or licensed
* Any condition requiring chronic use of steroids
* Any disorder with dysregulation of glucose homeostasis (history of Type 1 or 2 Diabetes Mellitus or prediabetic symptoms)
* History of glucose intolerance
* History of cetuximab infusion reactions
* Women of child-bearing potential unwilling or unable to use acceptable contraception methods

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of BMS-754807 administered orally (daily schedule) in combination with cetuximab administered standard doses IV (weekly basis) will be determined by observation of dose limiting toxicities during the first 33 days of administration | During and at the end of the first 33 days after the first dose of BMS-754807 is given

SECONDARY OUTCOMES:
To assess anti-tumor activity as measured by objective responses | every 8 weeks
To evaluate the safety and tolerability of the BMS-754807/cetuximab combination regimen | Ongoing
To assess the effects of the BMS-754807/cetuximab combination regimen on glucose homeostasis | Ongoing
Dose Expansion only: To identify biomarkers that are predictive of a response to BMS-754807/cetuximab combination therapy in advanced or metastatic CRC and SCCHN subjects with cetuximab resistance | tumor biopsies before treatment and on day 33 +/- 3 of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (5):
- United States (3):
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - University Of Wisconsin, Madison, Wisconsin
- Canada (2):
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Toronto, Ontario

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx